CLINICAL TRIAL: NCT02209350
Title: Prospective Randomized Clinical Study of the Aorto-femoral Bypass and the Iliac Arteries With Stenting Recanalization Effectiveness in Patients With the Iliac Segment Occlusive Disease
Brief Title: Study of the AFB and Stenting of the Iliac Arteries
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TASC C,D
Record Dates: First submitted 2014-07-30; First posted 2014-08-05 (Estimated); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Aorta-iliac Segment Lesion (C,D Type by TASC II)
MeSH Terms: interventions — Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Active Comparator): Operations technique on the abdominal aorta. Aorta-femoral bypass. Medication: after surgery all patients are prescribed long-term aspirin (100 mg daily) and clopidogrel for 3 months (75 mg daily).
  Interventions: Procedure: Aorta-femoral bypass; Drug: Therapy: aspirin and clopidogrel
- Group 2 (Active Comparator): Standard endovascular treatment (stenting) in patients with the iliac segment occlusive disease. Medication: after stenting all patients are prescribed long-term aspirin (100 mg daily) and clopidogrel for 3 months (75 mg daily).
  Interventions: Procedure: Recanalization and stenting of aorta-iliac segment; Drug: Therapy: aspirin and clopidogrel

INTERVENTIONS:
Procedure: Aorta-femoral bypass — Access to the femoral artery is performed through a lateral incision from the inguinal ligament. Operations technique on the abdominal aorta.
  Aorta-femoral bypass. Proximal anastomosis between the prosthesis and aorta is applied in the sort of "end-to-side" in the reconstruction by shunting.
  After jaws prosthesis conduction on hip distal anastomosis is formed with twisting controlling. In a case of preserved antegrade blood flow the femoral artery anastomosis applied in the sort of "end-to-side". If antegrade flow is absent, anastomosis is formed in the sort of "end to end".
  Arms: Group 1
Procedure: Recanalization and stenting of aorta-iliac segment — Standard endovascular access is performed under local anesthesia and affected arterial segment is visualized.
  Stenosis or artery occlusion is passed with hydrophilic guide. In case of occlusion transluminal or subintimal (often "mixed") artery recanalization is performed. To maximize the preservation of the affected artery initial patency, occlusion recanalization is performed by ante-and retrograde accesses. Then stenosis or occlusion predilation is performed with balloon catheter (balloon catheter diameter is smaller than the affected artery diameter for 1-2 mm). After control angiography stent is installed in the aorta-iliac area throughout the lesion (lesion diameter corresponds to the stenotic arteries diameter).
  Arms: Group 2
Drug: Therapy: aspirin and clopidogrel — prescribed long-term aspirin (100 mg daily) and clopidogrel for 3 months (75 mg daily).

SUMMARY:
The aim of the study is to compare effectiveness and long-term results of aorta-femoral reconstructions and endovascular treatment in the patients with aorta-iliac lesions (TASC C,D).

ELIGIBILITY:
Inclusion Criteria:

* Patients with unilateral steno-occlusive iliac lesions (TASC types C, D) and with chronic lower limb ischemia
* Rutherford classification category 3-5 chronic limb ischemia,
* age: 45-75 years old.
* Patients who consented to participate in this study.

Exclusion Criteria:

* Aortic thrombosis, concomitant abdominal aortic or iliac aneurysms, acute limb ischemia or vasculitis;
* Flush occlusion of the common iliac artery;
* Ipsilateral common femoral arteries steno-occlusive disease (occlusion or stenosis >50%);
* Ipsilateral profunda femoris artery steno-occlusive disease (occlusion or stenosis >50%);
* Refusal to participate in the study;
* Stroke or myocardial infarction within the past 3 months;
* Ischemic heart disease with New York Heart Association functional class IV;
* Malignant tumor with an estimated life span of under 6 months;
* Previous ipsilateral or contralateral surgery (bypass, hybrid or stenting);
* Hepatic or renal insufficiency (bilirubin> 35 mmol/l, glomerular filtration rate <60 ml/min/1.73 m2);
* Severe calcification of the aorta and iliac arteries intolerant to balloon angioplasty (as determined by the Peripheral Arterial Calcification Scoring System on computed tomography angiography as interpreted by a vascular radiologist):12
* unilateral calcification ≥ 5cm (Grade 2), bilateral calcification ≥ 5cm (Grade 4) or circumferential calcification , defined as 270°-360° around the circumference of aorta and/or iliac arteries.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2015-08-02 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2020-11-02 (Actual)

PRIMARY OUTCOMES:
Technical success | 1 day
  Successful implantation of all devices without the need for conversion and with residual stenosis less than 30%
30-day complication rate | 30 days
  clinically significant bleeding, hematoma, infection of the prosthesis, infection of postoperative wound, lymphorrhea, renal failure, myocardial infarction, stroke, mortality, thrombosis of the operated segment, distal embolism
30-day primary patency rates | 30 days
  during the whole 30 days from the date of intervention. confirmation of patency of the arterial ultrasound of the operated segment.
30-day secondary patency rates | 30-day
  during the whole 30 days from the date of intervention. confirmation of patency of the arterial ultrasound of the operated segment after reintervention due to thrombosis

SECONDARY OUTCOMES:
Major adverse cardiovascular event (MACE) | 36 months
  composite of nonfatal stroke, nonfatal myocardial infarction, and cardiovascular death
Limb salvage | 36 months
  preservation of a functional foot, eliminating the necessity for major amputation
Amputation-free survival | 36 months
  freedom from major limb amputation or death by any cause
Primary patency rates | 36 months
  no occlusion or significant flow-limiting stenosis in the treated segment
Secondary patency rates | 36 months
  no occlusion or flow-limiting stenosis following at least one re-intervention aimed at restoring patency, in addition to all instances of primary patency

CONTACTS AND LOCATIONS:
Overall Officials: Andrey Karpenko, MD, PhD, Principal Investigator — Novosibirsk Research Institute of Circulation Pathology
Locations (1):
- Novosibirsk Research Institute of Circulation Pathology, Novosibirsk, Russia